CLINICAL TRIAL: NCT06830018
Title: A Multicenter, Prospective, Randomized, Parallel-controlled Clinical Study of Nano-crystalline Megestrol Acetate Combined With Standard Treatment Versus Standard Treatment Alone for the First-line Treatment of Patients With Cancer-related Fatigue In Gastric Or Colorectal Cancer
Brief Title: Nanocrystalline Megestrol for First-line Treatment of Advanced Gastric or Colorectal Cancer With Cancer-related Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MGA- Fatigue-01
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Cancer-related Fatigue， Gastric Cancer，Colorectal Cancer，Nano-crystalline Megestrol Acetate，Megestrol Acetate，First-line Treatment
Keywords: cancer-related fatigue， cancer-caused fatigue，fatigue，appetite stimulants; gastric cancer，colorectal cancer，gastrointestinal tumor，cancer，tumor，carcinoma，; nano-crystalline megestrol acetate，megestrol，megestrol acetate，; antineoplastic agents, hormonal，central nervous system stimulants，appetite stimulants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-crystalline Megestrol Acetate Oral Suspension + Standard Therapy (Experimental)
  Interventions: Drug: Nano-crystalline Megestrol Acetate Oral Suspension; Combination Product: Standard Treatment
- Standard Therapy (Active Comparator)
  Interventions: Combination Product: Standard Treatment

INTERVENTIONS:
Drug: Nano-crystalline Megestrol Acetate Oral Suspension — Nano-crystalline Megestrol Acetate Oral Suspension, with a specification of 125 mg/mL, the study group takes 5 mL orally per day (625 mg/day), and continues medication; after completing the treatment cycle, patients who are assessed by the researchers as suitable for continued treatment may continue to receive therapy.
  Arms: Nano-crystalline Megestrol Acetate Oral Suspension + Standard Therapy
Combination Product: Standard Treatment — Standard Treatment，First-line treatment (chemotherapy + immunotherapy/targeted therapy)

SUMMARY:
This study is a prospective, randomized, parallel-controlled clinical trial, with the primary objective to evaluate the efficacy and safety of nano-crystalline megestrol acetate combined with standard treatment compared to standard treatment alone for the first-line treatment of patients with cancer-related fatigue in gastric or colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years.
* Eastern Cooperative Oncology Group (ECOG) physical status score of 0-2.
* Expected survival ≥ 6 months.
* Locally advanced or metastatic gastric/gastroesophageal junction (G/GEJ) adenocarcinoma or colorectal adenocarcinoma not amenable to radical treatment with histologic or cytologic confirmation.
* No prior systemic systemic antitumor therapy for gastric/gastroesophageal junction (G/GEJ) adenocarcinoma or colorectal cancer.
* Have at least one measurable tumor lesion according to RECIST v1.1.
* Compliance with a Fatigue Visual Analog Scale (VAS) score of ≥ 4 (consistent with moderate or severe fatigue).
* Complain of anorexia.
* Good organ function as determined by the following requirements.

Exclusion Criteria:

* Suffered significant surgery or traumatic injuries within the past 1month.
* Having any condition that affects gastrointestinal absorption, such as dysphagia, malabsorption, or uncontrollable vomiting.

currently undergoing tube feeding or parenteral nutrition.

* Suffering from anorexia due to neurosis, mental illness, or difficulty eating due to pain.
* Received erythropoietin or blood transfusion within the past 1month.
* Comorbidities such as serious cerebrovascular, heart, kidney, or liver disease.
* A history of hypersensitivity to the components of the trial medication.
* Other conditions that were considered inappropriate as determined by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
the difference in improvement of fatigue as measured with the Revised Piper Fatigue Scale-Chinese Version (RPFS-CV). | week 6
the difference in improvement of appetite based on A/CS-12 assessment | week 6

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital Of China Medical University, Shenyang, Liaoning, China